CLINICAL TRIAL: NCT03978624
Title: Window of Opportunity Platform Study to Define Immunogenomic Changes With Pembrolizumab Alone and in Rational Combinations in Muscle-Invasive Bladder Cancer
Brief Title: Window of Opportunity Study of Pembrolizumab Alone and in Combinations in Bladder Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCCC1827
Record Dates: First submitted 2019-04-22; First posted 2019-06-07 (Actual); Results first posted 2025-10-07 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Bladder Cancer
Keywords: Muscle Invasive Bladder Cancer; MIBC; pembrolizumab; entinostat
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — pembrolizumab; entinostat; Surgical Procedures, Operative; Cystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A: Pembrolizumab alone (Experimental): Subjects will be administered pembrolizumab alone 200 mg IV on day 1 and day 22
  Interventions: Drug: Pembrolizumab; Procedure: Procedure/Surgery
- B: Pembrolizumab plus Entinostat (Experimental): Subjects will be administered pembrolizumab on day 1 and day 22 and entinostat 5 mg given orally on day 1, day 8 and day 15
  Interventions: Drug: Pembrolizumab; Drug: Entinostat; Procedure: Procedure/Surgery

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg IV on day 1 and day 22
  Other Names: Keytruda
Drug: Entinostat — 5 mg given orally on day 1, day 8 and day 15
  Other Names: SNDX-275; MS-275
  Arms: B: Pembrolizumab plus Entinostat
Procedure: Procedure/Surgery — A radical cystectomy is a surgical procedure to remove the entire urinary bladder and maximal transurethral resection of bladder tumor (TURBT) is a surgical procedure used to remove as much of the bladder tumor as possible.
  Other Names: Radical cystectomy or maximal TURBT

SUMMARY:
This is an open-label, window of opportunity platform study for subjects with muscle-invasive bladder cancer (MIBC) who are deemed ineligible or refuse cisplatin-based neoadjuvant chemotherapy and are scheduled to undergo definitive surgery (radical cystectomy), or are planning to undergo trimodality therapy (maximal transurethral resection of the bladder tumor followed by concurrent chemoradiation).

The primary objective of this study is to assess changes to immunogenomic markers after treatment with pembrolizumab alone and in combination with the selective class I histone deacetylase (HDAC) inhibitor (entinostat).

DETAILED DESCRIPTION:
The study will enroll 20 subjects with a confirmed diagnosis of MIBC (cT2-T4aN0M0) who are planned for definitive therapy with either radical cystectomy without cisplatin-based neoadjuvant chemotherapy or trimodality therapy.

Prior to study entry, subjects must consent to having tissue collected for research purposes during the scheduled cystectomy or maximal TURBT. After screening and enrollment, baseline blood and archived transurethral resection of the bladder tumor (TURBT) tumor tissue will be collected from each subject for baseline analyses. Subjects will then start on clinical trial treatment followed by either radical cystectomy or maximal TURBT followed by chemoradiation.

Blood and tumor will be collected from each subject at the time of cystectomy or maximal TURBT. The investigators do not anticipate delays in surgery due to the planned schedule of the preoperative treatment administration for the purposes of this study and based on previous reported results of the trial which includes pembrolizumab and entinostat treatment in melanoma reported an acceptable safety profile. Phase I data identified grade 1/2 fatigue as the most common entinostat-related toxicity, with neutropenia and anemia only occurring at doses exceeding those proposed for this study. Safety stopping rules for drug-related toxicity will dictate whether the trial should be halted if subjects are experiencing drug-related toxicity that delays or interferes with the standard of care procedures.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained to participate in the study and HIPAA authorization for release of personal health information.
* Subjects must agree to donate tumor tissue from their transurethral resection of the bladder tumor (TURBT) and from their cystectomy, as well as agree to donate whole blood prior to initiating therapy, and at cystectomy.
* Age ≥18 years at the time of consent.
* Eastern Cooperative Oncology Group performance status of ≤ 2.
* Histological confirmation of urothelial carcinoma of the bladder; those with mixed histology, including a component of urothelial carcinoma, are eligible. Pure small cell carcinoma, pure adenocarcinoma, and pure squamous cell carcinoma are excluded.
* Subject has clinical stage T2-T4a N0/X M0 urothelial carcinoma. Clinical T stage is based on the pre-study standard of care transurethral resection of the bladder tumor (TURBT) sample and imaging studies (abdominal/pelvic CT or MRI scan and CT scan of the chest performed within 4 weeks prior to treatment initiation).
* Available formalin-fixed paraffin-embedded (FFPE) archival tumor specimen that contains sufficient tissue to generate at least 15 (preferably 20) unstained slides, each with tissue sections that are 5 - 10 microns thick.
* Subject is planned to undergo definitive surgery (radical cystectomy).
* Subject demonstrates adequate organ function as defined by the protocol; all screening laboratory assessments should be performed within 10 days of treatment initiation.
* Subject refuses to receive or is ineligible to receive cisplatin-based neoadjuvant chemotherapy. Determination of ineligibility for cisplatin is based on at least one of the following criteria:
* Eastern Cooperative Oncology Group performance status of 2
* Glomerular filtration rate (GFR) per Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation ≤ 60 mL/min
* NCI CTCAE v5.0 Grade ≥ 2 hearing loss
* NCI CTCAE v5.0 Grade ≥ 2 neuropathy
* Female subjects of childbearing potential should have a negative serum pregnancy within 72 hours prior to receiving the first dose of the study treatment.
* Female subjects of childbearing potential must be willing to use an adequate method of contraception as outlined in the protocol, for the course of the study through 120 days after the last dose of study medication.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

-Male subjects of childbearing potential must agree to use an adequate method of contraception as outlined in the protocol, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

* Subject is able to tolerate and retain oral medication.
* Life expectancy greater than 3 months.

Exclusion Criteria:

* Subject is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of pembrolizumab.
* Subject has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Inhaled and topical steroids are allowed.
* Subject has a known history of active tuberculosis.
* Subject has known hypersensitivity to pembrolizumab or any of its excipients.
* For subjects in arm 2 only, to benzamide or inactive ingredients of entinostat.
* Subject has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Subject has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Subject has a history of (non-infectious) pneumonitis that required steroids or a current pneumonitis.
* Subject has an active infection requiring systemic therapy.
* Subject has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator. Please note that subjects with Grade ≥2 peripheral neuropathy, are allowed on this study.
* Subject has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Subject is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Subject has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Subject has had prior systemic cytotoxic chemotherapy for urothelial carcinoma (prior intravesicular chemotherapies are permitted).
* Subject is receiving histone deacetylase inhibitors, including valproic acid, DNA methyltransferase inhibitors.
* For subjects in arm 2 only, subject is receiving drugs that are known to inhibit or induce P-gp.
* For subjects in arm 2 only, subject has gastrointestinal impairment that may significantly affect absorption of entinostat, such as ulcerative disease, malabsorption syndrome, and a history of small bowel resection.
* Subject has received prior radiation therapy to the bladder for the purpose of treating urothelial carcinoma.
* Subject has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Subject has known history of Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] has been detected).
* Subject has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
* For subjects in arm 2 only, subject uses drugs or herbal supplements that are known sensitive cytochromes P450 (CYP) substrates of CYP1A2, CYP2C8, CYP3A with narrow therapeutic range

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2026-11-22 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy L Rose, MD, Principal Investigator — UNC- Chapel HIll
Locations (2):
- United States (2):
  - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were enrolled in the study between 09/23/2020 and 04/18/2023 at two cancer centers in the United States.
Groups:
- Pembrolizumab: Patients will receive an infusion of pembrolizumab (200mg IV) on Day 1 and Day 22.
- Pembrolizumab Plus Entinostat: Patients will receive an infusion of pembrolizumab (200mg intravenous) on Day 1 and Day 22, as well as entinostat (50mg given orally) on Day 1, Day 8, and Day 15.
Period: Overall Study
Arm/Group | Pembrolizumab | Pembrolizumab Plus Entinostat
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants started the study activities.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab | Pembrolizumab Plus Entinostat | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Full Range); unit: years] | 73.5 [60 to 84] | 74.9 [62 to 86] | 74.2 [60 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 9 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 9 | 6 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Changes in CD8 T Cell Immune Gene Signature in the Pembrolizumab + Entinostat Group and the Pembrolizumab Group
Description: Gene expression levels with the CD8 T cell gene signature were measured using RNA sequencing. The expression level of each gene in the signature were log2 transformed and the mean of the signature genes was calculated in each sample. Then the mean expression of signature in each sample was compared to the average expression and variability across other sample to center the expression values (mean = 0) and scale them by standard deviation and generate a Z-score. Change in z-score was then calculated between pre- and post-treatments for each individual patient and then changes in z-score were compared between treatment arms. An increase in Z-score with treatment denotes an increase in expression of the immune gene signature (IGS).
Time Frame: Pre-treatment and at time of definitive treatment within 10 weeks after starting neoadjuvant treatment
Population: Participants started the study, and tissue analysis was completed.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Pembrolizumab | Pembrolizumab Plus Entinostat
Number analyzed (Participants) | 6 | 8
Z-score | 1.11 (1.39) | 1.01 (1.12)

2. Secondary Outcome: Change From Baseline in Number and Character of Neoantigens
Description: Neoantigens will be predicted based on whole exome sequencing data using mRNAseq-based filtering. The number of predicted neoantigens will be calculated in the pre-treatment biopsy specimen and the post-treatment cystectomy specimen for each patient. The change from baseline in number and character of neoantigens will be described and compared for each treatment group. Similarly, the T cell receptor (TCR) repertoire will be sequenced and clonality in blood and tumor will be compared between pre- and post-treatment samples for each patient, and change in clonality will be compared between treatment groups.
Time Frame: Less than 10 weeks
Reporting Status: Not Posted, anticipated posting 2027-11

3. Secondary Outcome: Change From Baseline in Signal Transducer and Activator of Transcription Factors (STAT) and Nuclear Factor Kappa-light-chain-enhancer of Activated B Cells (NF-κB) Gene Signatures and Histone Acetylation (H3K9Ac, H3K27Ac, and Others) Levels
Description: Compare changes in STAT and NF-κB gene signatures and histone acetylation (H3K9Ac, H3K27Ac, and others) levels after combination treatment with pembrolizumab and entinostat as compared to pembrolizumab alone (subset of subjects with frozen pre- and post-treatment tumor tissue available) Gene expression for each gene in representative STAT, NF-κB, and histone acetylation gene signatures (from MSigDB) will be quantified based on mRNA sequencing. Change in Z-score of these gene signatures will be calculated from pre- and post-treatment tissue samples for patients in both cohorts (pembrolizumab alone or pembrolizumab plus entinostat), and then changes in Z-scores will be compared between cohorts.
Time Frame: 10 weeks
Reporting Status: Not Posted, anticipated posting 2027-11

4. Secondary Outcome: Frequency and Severity of Attributed Adverse Events as Assessed by CTCAE v5.0
Description: The analysis of toxicity and safety will be based on the frequency and severity of adverse events attributed to the study treatment, occurring from Day 1 of treatment through 30 days after its completion. The worst toxicity grades per subject will be tabulated for adverse events and laboratory measurements using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v5.0) and reported in frequency tables.
Time Frame: 10 weeks
Population: Subjects started the treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Pembrolizumab Plus Entinostat
Number analyzed (Participants) | 10 | 10
Participants
  Grade 2 Hyperthyroidism | 1 | 0
  Grade 1 Diarrhea | 2 | 2
  Grade 1 Dry mouth | 1 | 0
  Grade 1 Nausea | 1 | 0
  Grade 1 Fatigue | 1 | 1
  Grade 1 Alanine aminotransferase increased | 1 | 0
  Grade 1 Alkaline phosphatase increased | 1 | 0
  Grade 1 Aspartate aminotransferase increased | 2 | 0
  Grade 1 Arthralgia | 1 | 0
  Grade 1 Myalgia | 0 | 1
  Grade 3 Myalgia | 1 | 0
  Grade 1 Pruritus | 1 | 0
  Grade 1 Rash maculo-papular | 1 | 0
  Grade 1 SFacial erythema/bilateral axilla rash | 1 | 0
  Grade 2 Skin tag | 0 | 1

5. Secondary Outcome: Proportion of Patients Who Have no Cancer in Tissue Samples at Surgery (Pathologic Complete Response, or Only Non-invasive Cancer (Pathologic Partial Response)
Description: The proportion of patients who have a pathologic response to less than stage 2 (<pT2) will be reported along with a 95% confidence interval. Similarly, the proportion of patients who have a complete response (pT0) will be reported.
Time Frame: 10 weeks
Population: Participants have started the study, completed surgery, and tumor response assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Pembrolizumab Plus Entinostat
Number analyzed (Participants) | 7 | 7
Participants
  Complete Response | 2 | 2
  Partial response / downstaging | 3 | 3

6. Secondary Outcome: Event Free Survival (EFS)
Description: EFS is defined as day 1 of neoadjuvant/protocol treatment to date of first documentation of disease progression (or until recurrence after surgery or radiation) or death due to any cause. Recurrence includes the development of second primary muscle-invasive urothelial malignancies.
Time Frame: Up to 3 years
Reporting Status: Not Posted, anticipated posting 2027-11

7. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as day 1 of neoadjuvant/protocol treatment to date of death due to any cause. Patients will be censored at date of last follow-up.
Time Frame: Up to 3 years
Reporting Status: Not Posted, anticipated posting 2027-11

ADVERSE EVENTS:
Time Frame: Up to 142 days of the last pembrolizumab administration.
Description: Adverse events were collected from day one of the study drug administration to 30 days after the last pembrolizumab administration according to National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE). All hospital admissions were graded as SAEs per protocol.
Arm/Group | A: Pembrolizumab Alone | B: Pembrolizumab Plus Entinostat
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 4/10 | 2/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A: Pembrolizumab Alone (N=10) | B: Pembrolizumab Plus Entinostat (N=10)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Confusion (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A: Pembrolizumab Alone (N=10) | B: Pembrolizumab Plus Entinostat (N=10)
Anemia (Blood and lymphatic system disorders) | 6 | 4
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 2 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 2 | 2
Diarrhea (Gastrointestinal disorders) | 4 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 1
Edema limbs (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 4
Vomiting (Gastrointestinal disorders) | 2 | 1
Fatigue (General disorders) | 4 | 2
Pain (General disorders) | 1 | 0
Rash pustular (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 4 | 2
Alanine aminotransferase increased (Investigations) | 2 | 1
Alkaline phosphatase increased (Investigations) | 2 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 1
Blood bicarbonate decreased (Investigations) | 1 | 0
Creatinine increased (Investigations) | 4 | 2
Lymphocyte count decreased (Investigations) | 1 | 2
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 4
Weight loss (Investigations) | 1 | 1
White blood cell decreased (Investigations) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 4
Hypokalemia (Metabolism and nutrition disorders) | 1 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 1
Proteinuria (Renal and urinary disorders) | 1 | 1
Urinary frequency (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Body odor (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 1
Hypertension (Vascular disorders) | 3 | 1
Hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Site shall not independently publish, present, or disclose the Study results, except as specified herein. If a joint publication is not submitted by the Institution within 18 months of the Study's conclusion, abandonment, or termination at all sites, the Site may publish. Additionally, the Site agrees to provide Syndax and Merck with a copy of any proposed publication at least 60 days before the intended publication date.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT03978624/Prot_SAP_000.pdf